CLINICAL TRIAL: NCT05433389
Title: App Delivered Brief Mindfulness Intervention for Knee or Hip Replacement Patients
Brief Title: App Delivered Brief Mindfulness Intervention for Surgical Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Adam Hanley, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00085446 AM_00032203
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Pain; Anxiety State; Depressive State
MeSH Terms: conditions — Pain; Anxiety Disorders; Depression | interventions — Whole Body Imaging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Breath Counting (Active Comparator)
  Interventions: Behavioral: Breath Counting
- Body Scan (Experimental)
  Interventions: Behavioral: Body Scan
- Mindful Breathing (Experimental)
  Interventions: Behavioral: Mindful Breathing
- Mindfulness of Pain (Experimental)
  Interventions: Behavioral: Mindfulness of Pain
- Mindful Savoring (Experimental)
  Interventions: Behavioral: Mindful Savoring

INTERVENTIONS:
Behavioral: Breath Counting — Patients will listen to a 5-minute, audio-recorded breath counting practice.
  Arms: Breath Counting
Behavioral: Body Scan — Patients will listen to a 5-minute, audio-recorded body scan practice.
  Arms: Body Scan
Behavioral: Mindful Breathing — Patients will listen to a 5-minute, audio-recorded mindful breathing practice.
  Arms: Mindful Breathing
Behavioral: Mindfulness of Pain — Patients will listen to a 5-minute, audio-recorded mindfulness of pain practice.
  Arms: Mindfulness of Pain
Behavioral: Mindful Savoring — Patients will listen to a 5-minute, audio-recorded mindful savoring practice.
  Arms: Mindful Savoring

SUMMARY:
This will be a single-site, five-arm, parallel group randomized control trial involving patients undergoing knee or hip replacement surgery. The investigators will compare five different styles of 5-minute, audio-recoded mindfulness practices delivered via app 7 days before to surgery, 2 days before to surgery, 2 days after surgery, and 6 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18,
* Scheduled to undergo total joint arthroplasty of the knee or hip

Exclusion Criteria:

* Inability to read English
* Cognitive impairment preventing completion of study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 823 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Unpleasantness | Immediately before to after 5-minute audio recording
  Single item assessing pain unpleasantness ("How unpleasant is your pain?") scored on an 11-point (0=Not at all, 10=Very much) numeric rating scale. Higher scores indicate greater pain unpleasantness.

SECONDARY OUTCOMES:
Change in Pain Intensity | Immediately before to after 5-minute audio recording
  Single item assessing pain intensity ("How much pain do you have?") scored on an 11-point (0=Not at all, 10=Very much) numeric rating scale. Higher scores indicate greater pain intensity.
Change in Pain Medication Desire | Immediately before to after 5-minute audio recording
  Single item assessing pain unpleasantness ("How much do you want pain medicine?") scored on an 11-point (0=Not at all, 10=Very much) numeric rating scale. Higher scores indicate greater desire for pain medicine.

OTHER OUTCOMES:
Change in Anxiety | Immediately before to after 5-minute audio recording
  Single item assessing pain unpleasantness ("How nervous, anxious, or on edge do you feel?") scored on an 11-point (0=Not at all, 10=Very much) numeric rating scale. Higher scores indicate greater anxiety.
Change in Depression | Immediately before to after 5-minute audio recording
  Single item assessing pain unpleasantness ("How down, depressed, or uninterested in life do you feel?") scored on an 11-point (0=Not at all, 10=Very much) numeric rating scale. Higher scores indicate greater depression.
Postoperative Patient Reported Outcomes Measurement Information System (PROMIS) Physical Functioning Item Bank, v2.0 | During the 6 weeks prior to surgery and at the 6-week outpatient follow-up appointment
  The PROMIS physical functioning computer assisted test draws from a bank of 123 items all scored on a 5 point Likert scale. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. A high score reflects better physical functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States